CLINICAL TRIAL: NCT00293176
Title: A One-Year, Multicenter, Randomized, Double-Blind, Placebo-Controlled Evaluation of the Efficacy and Safety of Donepezil Hydrochloride in Subjects With Mild Cognitive Impairment (MCI)
Brief Title: The Evaluation of the Efficacy and Safety of Donepezil Hydrochloride in Subjects With Mild Cognitive Impairment (MCI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-A001-412; NCT00100022 (obsolete NCT alias)
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Memory Loss
Keywords: Cognitive impairment; Memory Loss
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction | interventions — Donepezil

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Donepezil Hydrochloride
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil Hydrochloride — Subects will receive a starting dose of 5 mg orally. Dose-escalation from 5 mg to 10 mg will occur at the Week 9 Visit.
  Arms: 1
Drug: Placebo — Subjects will receive matching placebo tablets.
  Arms: 2

SUMMARY:
To investigate the efficacy and safety of donepezil in individuals with mild cognitive impairment on measures of cognition, global function and behavior.

ELIGIBILITY:
Inclusion Criteria:

* Memory complaint
* Mini Mental Status Exam (MMSE) score 24-28 inclusive
* General cognition and function performance sufficiently preserved such that a diagnosis of Alzheimer's disease (AD) cannot be made
* Generally healthy and ambulatory
* Sufficiently fluent in English

Exclusion Criteria:

* Diagnosis of probable or possible AD
* Neurological disorders
* History of malignant cancers
* Previously have taken donepezil or other acetylcholinesterase (ChE) inhibitors for more than 1 month or in the past 3 months prior to study entry

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 821 (Actual)
Dates: Start 2003-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Assessment of cognitive and global function in subjects with MCI.

SECONDARY OUTCOMES:
Behavioral, global and cognitive outcomes; Neuroimaging

CONTACTS AND LOCATIONS:
Overall Officials: Anita Murthy, Study Director — Eisai Inc.
Locations (54):
- United States (54):
  - Albaster, Alabama
  - Mesa, Arizona
  - Peoria, Arizona
  - Sun City, Arizona
  - Tucson, Arizona
  - Fresno, California
  - Garden Grove, California
  - Irvine, California
  - San Francisco, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Boynton Beach, Florida
  - Fort Meyers, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - North Miami, Florida
  - Ocala, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Venice, Florida
  - West Palm Beach, Florida
  - Snellville, Georgia
  - Chicago, Illinois
  - Elkhart, Indiana
  - New Orleans, Louisiana
  - Farmington Hills, Michigan
  - Kalamazoo, Michigan
  - Las Vegas, Nevada
  - Kenilworth, New Jersey
  - Long Branch, New Jersey
  - Albany, New York
  - Lexington, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - No. Charleston, North Carolina
  - Centerville, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Medford, Oregon
  - Portland, Oregon
  - Greensberg, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Madison, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Salt Lake City, Utah
  - Bennington, Vermont
  - Charlottesville, Virginia
  - Seattle, Washington